CLINICAL TRIAL: NCT01402817
Title: A Pilot Study of Sutent®/Sunitinib (SU11248), an Oral Multi-Targeted Tyrosine Kinase Inhibitor in Subjects With NF-1 Plexiform Neurofibromas
Brief Title: Study of Sutent®/Sunitinib (SU11248) in Subjects With NF-1 Plexiform Neurofibromas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 1 patient died of uncertain cause but possibly related to drug.
Sponsor: Indiana University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Pfizer (Industry)
Responsible Party: Principal Investigator, Chie-Schin Shih, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1104-07
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Neurofibromatosis; NF1; Plexiform Neurofibromas
Keywords: NF1; plexiform neurofibromas; Sunitinib; Sutent®
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma, Plexiform

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sutent®/Sunitinib (Experimental): Upon enrollment, subjects will receive Sutent® orally. Adults (Age >18) will receive 25mg. Children will receive 10mg/m2/day. All subjects will take the daily dose for 28 days followed by a 14 day rest period. If subjects tolerate the initial dose, adults will be increased to 37.5mg and children will be increased to 15mg/m2/day. Again, subjects will take that dose for 28 days followed by a rest period of 14 days. Adults who tolerate the increase will go up to the maximum dose of 50mg. The maximum dose for children is 15mg/m2/day.
  Interventions: Drug: Sutent®/Sunitinib

INTERVENTIONS:
Drug: Sutent®/Sunitinib — Upon enrollment, subjects will receive Sutent® orally. Adults (Age >18) will receive 25mg. Children will receive 10mg/m2/day. All subjects will take the daily dose for 28 days followed by a 14 day rest period. If subjects tolerate the initial dose, adults will be increased to 37.5mg and children will be increased to 15mg/m2/day. Again, subjects will take that dose for 28 days followed by a rest period of 14 days. Adults who tolerate the increase will go up to the maximum dose of 50mg. The maximum dose for children is 15mg/m2/day.

SUMMARY:
This is a pilot study to determine if adults and children with neurofibromatosis type 1 who have plexiform tumors given Sutent® respond to this drug therapy.

DETAILED DESCRIPTION:
This is an open-label pilot study to evaluate the efficacy of Sutent® in individuals with NF1 who have clinically significant plexiform tumors. A secondary goal of this study will be to seek to improve on current and novel tools to evaluate tumor response of plexiform tumors. The rationale for this study arises from the response of human and murine NF1 cells to Sutent® in vitro and the clinical response of individuals with NF1 using a similar drug,Gleevec®. Following enrollment adult subjects will start receiving Sutent® by month at 25mg once a day for 28 days. Subjects will then have 14 days without taking any Sutent®. If tolerated the dose will be increased to 37.5mg and 50mg with the same regimen (28 days of taking medication followed by 14 without). Children will be started on a dose of 10mg/m2/day once a day for 28 days. They will then have 14 days without taking any Sutent®. If tolerated the dose will be increased to 15mg/m2/day.

ELIGIBILITY:
Inclusion Criteria:

1. Age: patients must be ≥3 years of age and ≤65 years of age at the time of study entry
2. Diagnosis: Patients must meet clinical diagnostic criteria of neurofibromatosis type 1 (NF1). Patients must have clinically significant plexiform neurofibromas (biopsy proven if possible with tissue blocks available). Clinically significant tumors are those which are potentially life threatening or are impinging on vital structures or significantly impair the quality of life from pain or other symptoms.
3. Disease status: Patients must have measurable disease.
4. Performance Level: Karnofsky ≥50 for patients >10 years of age and Lansky ≥50 for patients ≤10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Prior therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

   1. Myelosuppressive chemotherapy: Must not have received within 3 weeks of entry onto this study.
   2. Hematopoietic growth factors: At least 14 days since completion of therapy with a growth factor.
   3. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, the period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the principal investigator.
   4. XRT: ≥2 weeks for local palliative XRT (small port); ≥6 months must have elapsed if ≥50% radiation of pelvis; ≥6 weeks must have elapsed if other substantial BM radiation.
6. Organ function requirements

   a. Adequate bone marrow function defined as i. Peripheral absolute neutrophil count (ANC) ≥1000/µL ii. Platelet count ≥100,000/ µL(transfusion independent, iii. Hemoglobin ≥8.0 gm/dL(may receive RBC transfusions) b. Adequate renal function defined as i. Creatinine clearance or radioisotope GFR ≥70 mL/min/1.73 m2 or ii. A serum creatinine based on age/gender as follows (Maximum Serum Creatinine (mg/dL)): Males: 6 to <10 years:1; 10 to <13 years: 1.2; 13 to <16 years: 1.5; >16 years 1.7. Females: 6 to <10 years:1; 10 to <13 years 1.2; 13 to <16 years: 1.4; >16 years: 1.4.

   The threshold creatinine values above were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

   c. Adequate Liver Function Defined As: i. Total bilirubin (sum of conjugated+unconjugated)≤1.5 times upper limit of normal (ULN) for age, and ii. SGPT(ALT)<2.5 upper limit of normal ULN). For the purpose of this study, the ULN for SGPT is 45 U/L iii. Serum albumin ≥2 g/dL d. Adequate cardiac function defined as: i. Shortening fraction or ejection fraction greater than the LLN (institutional norm), and ii. Corrected QT interval ≤450 msec e. Normal Pancreatic function defined as: i. Serum amylase ≤1.5xULN and ii. Serum lipase ≤1.5xULN. f. Blood pressure within the upper limit of normal defined as: i. A blood pressure (BP) ≤ 95th percentile for age, height, and gender and not receiving medication for treatment of hypertension.
7. Informed Consent: All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

   -

Exclusion Criteria:

1. Prior anthracycline treatment. Patients previously treated with anthracyclines (any dose) are not eligible.
2. Prior Cardiac Radiation Patients previously treated with a radiation field that included the heart are not eligible.
3. Pregnancy or Breast-Feeding Animal studies indicate an increased risk of death of pregnant female rats and rabbits exposed to Sutent®. Cleft lip and palate were observed in some fetuses exposed in utero to sunitinib. There is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are poet-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
4. Concomitant Medications

   1. Growth factors(s): Growth factors that support platelet or white cell number or function must not have been administered within the past 14 days
   2. Investigational Drugs: Patients who are currently receiving another investigational drug.
   3. Anti-cancer agents: Patients who are currently receiving other anti-cancer agents.
   4. The following CYP3A4 inducers are prohibited 12 days before the start of Sutent® and during the study with Sutent®: rifampin, rifabutin, carbamazepine, Phenobarbital, phenytoin, St. John's wort, efavirenz, and tipranavir.
   5. Anti-thrombotic and anti-platelet agents: warfarin (Coumadin), heparin, low molecular weight heparin, aspirin, and/or ibuprofen, or other NSAIDs.
   6. The following CYP3A4 inhibitors are prohibited 7 days before the start of sunitinib and during the study with sunitinib: azole antifungals (itraconazole, ketoconazole); clarithromycin, erythromycin, diltiazem, verapamil, HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir); delavirdine.
5. Infection: Patients who have an uncontrolled infection.
6. Pleural-based tumors: Pediatric patients treated on a phase II trial with imatinib had a higher than expected rate of hemorrhagic pleural effusions. Sutent® inhibits two of the same receptor tyrosine kinases as imatinib, PDGFR and c-KIT. Patients with tumors involving or abutting the pleural surface will be excluded from study. Patients with pulmonary lesions should be monitored closely for the development of hemorrhagic pleural effusions.
7. Patient size: Due to dosing limitations, patients with body surface area <0.5 m2 will be excluded from study.
8. Patients with a pre-existing thyroid abnormality (hyper-or hypothyroidism) with unstable thyroid function will be excluded from study. For the purposes of this study, unstable thyroid function will be defined as thyroid function abnormalities requiring more than on e change in thyroid medication in the 6 months prior to study entry.
9. Patients with history of allergic reaction attributed to Sutent® or component of Sutent® capsules.
10. Prior use of Sutent®: Patients who have previously received sunitinib are not eligible for study.
11. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
12. Patient is < 5 years free of another primary malignancy except if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
13. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
14. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
15. Patient has a known brain metastasis. Non-specific CNS changes on MRI/CT characteristic of NF1 are allowed, but not known CNS malignancies.
16. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
17. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
18. Patient had a major surgery within 2 weeks prior to study entry.

    -

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chie-Schin Shih, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sutent®/Sunitinib: Upon enrollment, subjects will receive Sutent® orally. Adults (Age >18) will receive 25mg. Children will receive 10mg/m2/day. All subjects will take the daily dose for 28 days followed by a 14 day rest period. If subjects tolerate the initial dose, adults will be increased to 37.5mg and children will be increased to 15mg/m2/day. Again, subjects will take that dose for 28 days followed by a rest period of 14 days. Adults who tolerate the increase will go up to the maximum dose of 50mg.The maximum dose for children is 15mg/m2/day.
Period: Overall Study
Arm/Group | Sutent®/Sunitinib
Started | 19
Completed | 8
Not Completed | 11
Not completed — Withdrawal by Subject | 3
Not completed — Study Suspended by FDA | 8

BASELINE CHARACTERISTICS:
Arm/Group | Sutent®/Sunitinib
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: To estimate the disease control rate (SD, PR, CR) with Sutent® in patients with neurofibromas (NF1). Tumor response criteria are determined by changes in size using all 3 dimensional measurements: width (W), transvers (T) , and length (L) measurements. Partial Response: ≥20% decrease in the sum of the products of the three perpendicular diameters of all target lesions (up to 5), taking as reference the initial baseline measurements.Stable Disease (SD): Neither sufficient decrease in the sum of the products of the three perpendicular diameters of all target lesions to qualify for PR (taking as reference the initial baseline measurements), nor sufficient increase in a single target lesions to qualify for PD, (taking as reference the smallest disease measurement since the treatment started).Progressive Disease (PD): 40% or more increase in the product of perpendicular diameters of ANY target lesion, taking as reference the smallest product observed.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Sutent®/Sunitinib: Upon enrollment, subjects will receive Sutent® orally. Adults (Age >18) will receive 25mg. Children will receive 10mg/m2/day. All subjects will take the daily dose for 28 days followed by a 14 day rest period. If subjects tolerate the initial dose, adults will be increased to 37.5mg and children will be increased to 15mg/m2/day. Adults who tolerate the increase will go up to the maximum dose of 50mg. The maximum dose for children is 15mg/m2/day.
Arm/Group | Sutent®/Sunitinib
Number analyzed (Participants) | 19
percentage of subjects | 52 [39.21 to 77.73]

2. Secondary Outcome: Volumetric Disease Evaluation
Description: To determine the response rate with Sutent® in patients with plexiform neurofibromas using volumetric analysis of MRI scans
Time Frame: 6 months
Measure: Number; unit: percentage of subjects
Arm/Group | Sutent®/Sunitinib
Number analyzed (Participants) | 19
percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the time subjects were taking drug and 30 days following completion of therapy
Arm/Group | Sutent®/Sunitinib
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sutent®/Sunitinib (N=19)
seizure (Nervous system disorders) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sutent®/Sunitinib (N=19)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
alanine aminotransferase increased (Investigations) | 1 (2)
alkaline phosphatase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
blood bilirubin increased (Investigations) | 3 (4)
cognitive disturbance (Nervous system disorders) | 1 (2)
chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
depression (Psychiatric disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
Hypercalcemia (Investigations) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hyperuricemia (Investigations) | 2 (4)
Hypoalbuminemia (Investigations) | 1 (1)
hypocalcemia (Investigations) | 1 (1)
hypokalemia (Investigations) | 1 (1)
Hpomagnesemia (Investigations) | 1 (1)
Hypophoshatemia (Investigations) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
neutrophil count decreased (Investigations) | 9 (11)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pain (General disorders) | 4 (4)
palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
pain in extremity (General disorders) | 1 (1)
platelet count decreased (Blood and lymphatic system disorders) | 5 (5)
Rash aceniform (Skin and subcutaneous tissue disorders) | 1 (1)
scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
serum amylase increased (Investigations) | 2 (3)
sinusitis (Infections and infestations) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (3)
vomiting (Gastrointestinal disorders) | 2 (3)
white blood cell decreased (Investigations) | 13 (13)
generalized muscle weakness (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes